CLINICAL TRIAL: NCT02101970
Title: Randomized Pilot Trial of Omega-3 Fatty Acids or Placebo in Peri- or Post-Menopausal Women at High Risk for Breast Cancer Undergoing a Weight Loss Intervention
Brief Title: Weight Loss Plus Omega-3 Fatty Acids or Placebo in High Risk Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00000703
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer
Keywords: Breast cancer risk; DHA; Omega-3 Fatty Acids; EPA; Weight Loss
MeSH Terms: conditions — Breast Neoplasms; Weight Loss | interventions — Fatty Acids, Omega-3; Eicosapentaenoic Acid; Docosahexaenoic Acids; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weight Loss + Omega-3 FA (Experimental): Participants will be instructed to follow a diet that is reduced by 500-700 kcal/day below maintenance requirements for 24 weeks or until the individual has reached a BMI of 25kg/m2 (generally 1000-2000 calories/day). Participants will be given one capsule of Omega-3 FA (fatty acids) a day beginning 2 weeks after starting their diet and exercise routine. Omega-3 FA will be increased by 1 capsule/day or every other day until participant is taking 5 capsules per day.Each Amber 4020 Ethyl Ester (EE) 1000 mg omega-3 capsule contains 420 mg of EPA and 210 mg of DHA both as the ethyl esters (380 mg EPA and 190 mg DHA)
  Interventions: Dietary Supplement: Omega-3 Fatty Acids; Other: Diet and Exercise
- Weight Loss + Placebo (Active Comparator): Participants will be instructed to exercise and follow a diet that is reduced by 500-700 kcal/day below maintenance requirements for 24 weeks or until the individual has reached a BMI of 25kg/m2 (generally 1000-2000 calories/day). Participants will be given one capsule of placebo a day beginning 2 weeks after starting their diet and exercise routine. Placebo capsule will be increased by 1 capsule/day or every other day until participant is taking 5 capsules per day.
  Interventions: Other: Placebo Capsule; Other: Diet and Exercise

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids — Amber 4020 Ethyl Ester (EE) 1000 mg omega-3 capsule contains 420 mg of EPA and 210 mg of DHA both as the ethyl esters (380 mg EPA and 190 mg DHA)
  Other Names: Eicosapentaenoic Acid (EPA); Docosahexaenoic Acid (DHA)
  Arms: Weight Loss + Omega-3 FA
Other: Placebo Capsule
  Arms: Weight Loss + Placebo
Other: Diet and Exercise — Increasing physical activity required over 6 month period to be tracked by a Fitbit. Diet based on caloric intake and eating approved foods.

SUMMARY:
The purpose of this study is to determine if high dose supplementation with the omega-3 fatty acids EPA and DHA, when added to a weight loss program, is well tolerated in the study population and if there is an increase in the favorable change in blood and tissue breast cancer risk factors when compared to weight loss alone.

DETAILED DESCRIPTION:
Subjects will all participate in a 6-month weight loss intervention. Subjects will be randomized to receive either blinded placebo or omega-3 fatty acids for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of Hyperplasia with Masood score of 13 or higher and 500 or more epithelial cells on cytology slide of screening Random Periareolar Fine Needle Aspiration (RPFNA)
* Access to smart phone and or computer
* Willing to comply with diet, exercise and lifestyle modification during weight reduction and maintenance phase.
* Willing to start the dietary and exercise intervention within 9 months of RPFNA
* Willing to complete quality of life questionnaires at multiple visits
* Willing to have a medical history and physical at multiple visits
* Willing to have an additional RPFNA at two additional visits
* Be willing to have blood drawn at multiple visits
* Willing to sign and able to understand consent for the RPFNA's and study participation
* Reasonable hematopoetic, kidney and liver function consistent with safe participation on this trial.

Exclusion Criteria:

* Having taken medications that seriously affect metabolism such as steroids, dexatrim or other diet drugs within 3 weeks of study registration
* Have changed dose or type of hormone supplementation within 3 months
* Currently receiving other investigational agents
* Have been on a chemoprevention trial within 6 months or taken a Selective Estrogen Receptor Modulator or aromatase inhibitor within last 6 months.
* Need for chronic use of aspirin, nonsteroidal anti-inflamatory drug (NSAID) or other anti-inflammatory agents
* Taking metformin, or other diabetes medications
* Taking statins
* Unable to participate in moderate intensity exercise (walking, treadmill, elliptical, water aerobics)
* Would be unable to participate, by phone, in weekly phone call sessions
* Cells suspicious for malignancy as assessed by cytotechnologist or cytopathologist.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2018-08-27 (Actual)

PRIMARY OUTCOMES:
Dropout rate | Up to 6 Months
  Measured as the number of participants that dropout before diet+intervention period is complete

SECONDARY OUTCOMES:
Study design feasibility | Up to 6 months
  Based on eligibility criteria, study procedures and participation of subjects the study design will be measured to see if it will practically work with a larger study population
Modulation of breast cancer risk biomarkers | Change from Baseline to 6 Months
  Measure the change in fasting and postprandial blood inflammatory, and risk biomarkers
Modulation of breast cancer risk biomarkers in benign breast tissue | Change from Baseline to 6 Months
  Measure change in fasting and postprandial blood inflammatory, and risk biomarkers
Modulation of breast cancer risk biomarkers | Change from Baseline to 12 Months
  Measure the change in fasting and postprandial blood inflammatory, and risk biomarkers
Modulation of breast cancer risk biomarkers in benign breast tissue | Change from Baseline to 12 Months
  Measure change in fasting and postprandial blood inflammatory, and risk biomarkers
Weight gain | Change from 6 Months to 12 Months
  Measure change in weight in participants during the 6-12 month maintenance phase
Change in Gut Microbiome | Change from Baseline to Month 6
  Change in eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA):arachidonic acid (AA) ratio

CONTACTS AND LOCATIONS:
Overall Officials: Carol J. Fabian, M.D., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Breast Cancer Prevention Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No
Global results will be published.

REFERENCES:
- [Result] Fabian CJ, Befort CA, Phillips TA, Nydegger JL, Kreutzjans AL, Powers KR, Metheny T, Klemp JR, Carlson SE, Sullivan DK, Zalles CM, Giles ED, Hursting SD, Hu J, Kimler BF. Change in Blood and Benign Breast Biomarkers in Women Undergoing a Weight-Loss Intervention Randomized to High-Dose omega-3 Fatty Acids versus Placebo. Cancer Prev Res (Phila). 2021 Sep;14(9):893-904. doi: 10.1158/1940-6207.CAPR-20-0656. Epub 2021 Jul 9. PMID 34244155